CLINICAL TRIAL: NCT03847818
Title: A Prospective, Open-label,Multicenter Phase II Study of Neoadjuvant Pyrotinib Plus Trastuzumab and Chemotherapy in Women With HER2 Positive Early Stage or Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Study of Pyrotinib and Trastuzumab Plus Chemotherapy in Patients With HER2 Positive Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yu-Zhi Gang, Director, The Second Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 495573096
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: Pyrotinib (400mg orally daily)+Trastuzumab (8mg/kg iv load followed by 6mg/kg iv 3-weekly)+Docetaxel (75mg/m2)+ Carboplatin(AUC=5/6), for a total of 4 cycles.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib+Trastuzumab+Docetaxel+Carboplatin (Experimental)
  Interventions: Drug: Pyrotinib+Trastuzumab+Docetaxel+Carboplatin

INTERVENTIONS:
Drug: Pyrotinib+Trastuzumab+Docetaxel+Carboplatin — Drug: Pyrotinib Pyrotinib: 400mg orally daily
  Drug: Trastuzumab Trastuzumab:8mg/kg iv load followed by 6mg/kg iv 3-weekly for a total of 6 cycles;
  Drug: Docetaxel Docetaxel: 75mg/m2 for a total of 6 cycles
  Drug: Carboplatin Carboplatin: AUC=5 or 6 for a total of 6 cycles

SUMMARY:
This is a prospective, open-label,multicenter Phase II study for evaluating the efficacy and safety of neoadjuvant pyrotinib and trastuzumab plus chemotherapy as neoadjuvant treatment in HER2 positive early stage or locally advanced breast cancer.

DETAILED DESCRIPTION:
The investigators hypothesized that the experimental group (Pyrotinib+Trastuzumab+Docetaxel+ Carboplatin) could have a higher Pathological Complete Response (pCR) rate than the control group (Trastuzumab+Docetaxel+ Carboplatin) in neoadjuvant chemotherapy.

It is proposed that 268 participants will be enrolled in this study. The target population is women with early breast cancer (stage of T2-3N0-3M0) who are eligible for primary systemic therapy.

The primary objective of the trial is to determine the pCR rate. The secondary objective of the trial is to determine the Event-free survival(EFS), Disease-free Survival (DFS), Distance Disease-free Survival (DDFS), Objective Response Rate (ORR) rate.

ELIGIBILITY:
Inclusion Criteria:

1. female patients, 18 years ≤ age ≤75 years；
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1;
3. Histologically confirmed invasive breast cancer（early stage or locally advanced）
4. HER2 positive (HER2+++ by IHC or FISH+)
5. Known hormone receptor status.
6. Cardiovascular: Baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO
7. Signed informed consent form (ICF)

Exclusion Criteria:

1. Metastatic disease (Stage IV) or inflammatory breast cancer.
2. Previous or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin, Carcinoma in situ of the cervix.
3. Clinically relevant cardiovascular disease: Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
4. Unable or unwilling to swallow tablets.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Event-free survival | Following surgery until Year 3
Disease-free Survival | Following surgery until Year 3
Distance Disease-free Survival | Following surgery until Year 3
Objective Response Rate | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery) up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhigang, DR., Principal Investigator — The Second Hospital of Shandong University